CLINICAL TRIAL: NCT03498443
Title: Effect of Pelvic Organ Prolapse Surgeries on Female Sexual Function in Egyptian Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Ashraf samir MD, lecturer of obstetrics and gynecology BeniSuef university, Beni-Suef University
Other Study IDs: Asamir
Record Dates: First submitted 2018-04-08; First posted 2018-04-13 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Female Sexual Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
study on female sexual function after different prolapse surgeries

ELIGIBILITY:
Inclusion Criteria:

* sex active prolapse surgery

Exclusion Criteria:

* not sex active any psychiatric problem

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: females e prolapse ser
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-05-01 (Estimated)

PRIMARY OUTCOMES:
sexual function after prolapse surgeries | month3
  questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Benisuef Uneversity Hospital, Banī Suwayf, BeniSuef, Egypt